CLINICAL TRIAL: NCT07218237
Title: Mindfulness and Wearable Biosensors to Prevent Hypertensive Disorders of Pregnancy Study: MINDBP
Brief Title: Mindfulness and Wearable Biosensors to Prevent Hypertensive Disorders of Pregnancy
Acronym: MINDBP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Anna Palatnik, MD, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO00056473
Record Dates: First submitted 2025-09-18; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Preeclampsia
Keywords: Hypertensive disorders of pregnancy; Mindfulness; Biofeedback
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Who Masked: Participant
Masking Description: All participants will wear a Garmin Vivoactive 4 biosensor watch throughout the study. However, only one of the arms will have real-time access to thier data, while the other 2 arms will be masked to their watch data. The study team will have access to the watch data for all 3 arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MT + Biofeedback (Experimental): Mindfulness training plus self-monitoring with access to data from wearable biosensor
  Interventions: Behavioral: Mindfulness training; Behavioral: Garmin Vivoactive 4 watch
- MT (Experimental): Mindfulness training (no access to wearable biosensor data)
  Interventions: Behavioral: Mindfulness training
- Control (No Intervention): Routine prenatal care alone

INTERVENTIONS:
Behavioral: Mindfulness training — Mindfulness training with trained instructors
  Arms: MT; MT + Biofeedback
Behavioral: Garmin Vivoactive 4 watch — Biofeedback with a wearable biosensor that continuously monitors heart rate variability and generates stress scores.
  Arms: MT + Biofeedback

SUMMARY:
The MINDBP study will enroll 90 pregnant women at risk for HDP across two sites (MCW and Brown) and randomize them to: (1) mindfulness training (MT) plus wearable biosensors, (2) MT alone, or (3) routine prenatal care. MT participants will receive 8 weekly phone-based MT sessions plus two booster sessions at 1 and 2 months post-intervention. The primary outcome is study feasibility.

DETAILED DESCRIPTION:
The MINDBP study will enroll 90 pregnant women at risk for HDP across two sites (MCW and Brown) and randomize them to: (1) MT + wearable biosensors, (2) MT alone, or (3) routine prenatal care. MT participants will receive 8 weekly phone-based MT sessions plus two booster sessions at 1 and 2 months post-intervention. All participants will wear Garmin Vivoactive 4 watches. Blood pressure, heart rate, heart rate variability, perceived stress, and pregnancy-related anxiety will be assessed at baseline (≤16 weeks), post-intervention (~24 weeks), and after each booster (~28 and 32 weeks). Feasibility, fidelity, and acceptability outcomes will be assessed after each post-intervention

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients at gestational age <= 16 weeks
* Live, non-anomalous gestation
* Normotensive at enrollment
* Meet criteria consistent with 'moderate' to 'high' risk for preeclampsia based on ACOG/USPSTF guidelines for low-dose aspirin administration to prevent hypertensive disorders of pregnancy

Exclusion Criteria:

* Multiple gestation
* Chronic (pregestational hypertension)
* Inability of unwillingness to provide informed consent
* Active suicidality or psychosis
* Ongoing mind-body practice (e.g., yoga, meditation, mindfulness >= once per week)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of multisite RCT | 3 years
  Assess study feasibility as measured by retention rate

SECONDARY OUTCOMES:
Acceptability of MINDBP intervention | Collected at the 3 study visits: 1 week, 1 month, and 2 months after completion of 8-week mindfulness training intervention.
  Assess intervention acceptability using Theoretical Framework of Acceptability Questionns (TFAQ). The TFAQ include 8 Likert-scale items which are averaged to provide an overall score from 1-5, with 5 indicating higher acceptability.
Home blood pressure | Daily blood pressure measurements for 6 weeks throughout the study
  Average systolic and diastolic blood pressure measured using home blood pressure monitoring
Heart rate variability | Up to 34 weeks
  Average daily stress score based on heart rate variability from biosensor watch
Perceived stress | Measured at baseline and 2, 3, and 4 months after consent.
  Self-reported perceived stress using the Perceived Stress Scale, which is scored from 0-40, with higher scores indicating higher perceived stress.
Pregnancy-related anxiety | Measured at baseline and 2, 3, and 4 months after consent.
  Self-reported pregnancy-related anxiety using the PRAQ-R2, which is cored from 0-40, with higher scores indicating higher anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Palatnik, MD, Principal Investigator — Medical College of Wisconsin; Margaret Bublitz, PhD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Brown University, Providence, Rhode Island
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Data collected in the study will include information collected from participants during pregnancy and up to 6 weeks postpartum. Variables will include demographic information, participant-reported survey data, wearable biosensor data, and maternal blood pressure from n=90 participants. All data will be de-identified prior to data sharing.
Supporting Information: Study Protocol, ICF
Time Frame: The repository will make the data accessible within 2 years of the last patient's last study visit or at the end of the performance period, or no later than the date of publication, whichever is sooner. Data will be preserved within the repositories for at least three years following the completion of the grant, as required by federal retention guidelines.
Access Criteria: Data that are necessary for and of sufficient quality to validate and replicate the study findings for the primary aims will be shared. We agree that the data will be deposited and made available as public use data to the research community via BioLINCC, and that these data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA) and can be used for secondary study purposes. We agree that the names and institutions of persons either given or denied access to the data, and the basis for such decisions, will be summarized in the annual progress report. Interested investigators will need to seek approval for data access from the contact PI.